CLINICAL TRIAL: NCT05466526
Title: Microinvasive Glaucoma Surgery -The Lowering Effect of Intraocular Pressure on Glaucoma Patients With High Frequency Deep Sclerotomy
Acronym: HFDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: Local clinic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-042-F
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Primary Open Angle Glaucoma; Intraocular Pressure; Glaucoma Surgery
Keywords: Primary Open Angle Glaucoma; High frequency deep sclerotomy; Abee glaucoma tip of Oertli
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: All participants in the arm were suffering from chronic open-angle glaucoma and were indicated for surgery due to either progression of field defect and raised intraocular pressure above 21 mmHg in spite of maximum medical treatment or for patients who were not compliant patient to their medical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The participants who received HFDS (Experimental): All participants in the arm were suffering from primary open-angle glaucoma and were indicated for surgery due to either progression of field defect and raised intraocular pressure above 21 mmHg in spite of maximum medical treatment or for patients who were not compliant patient to their medical treatment.
  Interventions: Procedure: High frequency deep sclerotomy (HFDS)

INTERVENTIONS:
Procedure: High frequency deep sclerotomy (HFDS) — The surgery was performed using the abee® glaucoma tip of Oertli phacoemulsiﬁcation machine (Cata-rhex3, Switzerland) and goniolens. During the procedures, nasal six pockets penetrating 1mm deep from the trabecular meshwork to Schlemm's canal will be formed to promote the aqueous humor outflow.

SUMMARY:
Highlights the high-frequency deep sclerotomy (HFDS) as a promising ab-interno surgery in primary open-angle glaucoma (POAG) patients and evaluates the eﬃcacy and safety of the procedure.

DETAILED DESCRIPTION:
[Materials and Methods ] This is a single-centre, prospective, non-blinded, interventional trials designed to evaluate the therapeutic effect and safety of HFDS in POAG patients. A total of 30 subjects were recruited, all of whom were outpatients of the ophthalmology department of attending physician MeiLan Ko in the National Taiwan University Hospital Hsin-Chu Branch. The 20 subjects were all diagnosed with POAG. The surgery was performed in the surgery room of the National Taiwan University Hospital Hsin-Chu Branch. The surgery was performed using the abee® glaucoma tip of Oertli phacoemulsiﬁcation machine (Cata-rhex3, Switzerland) and goniolens. During the procedure, nasal six pockets penetrating 1mm deep into the trabecular meshwork and Schlemm's canal were formed to promote aqueous humor outflow.

[Postoperative follow-up and evaluation] The postoperative IOP and visual acuity (VA) were measured in every follow-up visit for 6 months. Postoperatively, Cravit/Lotemax drops were given to prevent inflammation and infections; besides, Pilocarpine 2% eye drops were provided to reduce IOP for postoperative medication.

[Data Statistics and Analysis] Statistical analysis was done by IBMSPSS v21.0 statistical software (IBM Corporation, New York, USA). Data analysis was done by chi square (χ2) test, paired samples T-test and repeated ANOVA measurements with Bonferroni post hoc analysis. The results are considered statistically signiﬁcant with a P value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic open angle glaucoma and were indicated for surgery due to either progression of field defect and raised intraocular pressure above 21 mmHg in spite of maximum medical treatment or for patients who were not compliant patient to their medical treatment.

Exclusion Criteria:

* Patients with close-angle, congenital, traumatic, neovascular, and uveitic glaucoma, patients with prior penetrating and nonpenetrating glaucoma surgeries or laser therapy, and eyes with corneal opacity precluding visualization of the angle.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of intraocular pressure (IOP) after HFDS treatments compared to preoperative IOP. | Postoperative day 1, day 7, day 14, 1st month, 2nd month, 3rd months, 4th month, 5th month and 6th months.
  The postoperative IOP will be measured in every follow-up visit for 6 months after the operation. If the IOP of the participants is lower than that before the operation, and there is no tendency to increase within six months as well as no additional complications occur, the benefits of the primary outcome will be achieved.

SECONDARY OUTCOMES:
Change of visual acuity (VA) after HFDS treatments compared to preoperative VA. | Postoperative day 1, day 7, day 14, 1st month, 2nd month, 3rd months, 4th month, 5th month and 6th months.
  The postoperative visual acuity(VA) will be measured in every follow-up visit for 6 months after the operation. If the VA of the participants is getting better than that before the operation, and there is no tendency to worse within six months as well as no additional complications occur, the benefits of the secondary outcome will be achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Li Min-Zhen, investigator, Principal Investigator — IRB of NTUH Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report (CSR) can be shared
Supporting Information: CSR
Time Frame: After clinical study report (CSR) are posted; No definite time frame
Access Criteria: No limit